CLINICAL TRIAL: NCT01754194
Title: An Observational Study in Morbidly Obese Patients to Evaluate Laparoscopic Gastric Sleeve Resections and Roux-en-Y Gastric Bypass Surgery in Clinical and Health-Economic Terms
Brief Title: Clinical and Economic Outcomes in Laparoscopic Sleeve Gastrectomy Versus Roux-en-Y Gastric Bypass Surgery
Acronym: OPTIMIZE
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVMBSG0167
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Results first posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-04

CONDITIONS: Morbid Obesity
Keywords: Gastric Sleeve; Gastric Bypass; Roux en Y; Morbid Obesity; Laparoscopy
MeSH Terms: conditions — Obesity, Morbid | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Procedure Type 1: Gastric Sleeve Resection
  Interventions: Procedure: Gastric Sleeve Resection
- Procedure Type 2: Roux-en-Y Gastric Bypass
  Interventions: Procedure: Roux-en-Y Gastric Bypass

INTERVENTIONS:
Procedure: Gastric Sleeve Resection — Laparoscopic Gastric Sleeve Resection
  Groups: Procedure Type 1
Procedure: Roux-en-Y Gastric Bypass — Laparoscopic Roux-en-Y Gastric Bypass
  Groups: Procedure Type 2

SUMMARY:
Study objectives:

1. generate local clinical, health-related quality-of-life and health economic data to evaluate the benefits of two types of minimally invasive weight-loss surgery
2. support multi-disciplinary bariatric sites in Germany by providing structured procedure guidelines and training, therefore facilitating procedural adoption, increasing safety and shortening the learning curve for weight-loss surgery.

DETAILED DESCRIPTION:
The objectives of this study are the following: to generate local clinical, health-related quality-of-life and health economic data to evaluate the benefits of two types of minimally invasive weight-loss surgery; and to support multi-disciplinary bariatric sites in Germany by providing structured procedure guidelines and training, therefore facilitating procedural adoption, increasing safety and shortening the learning curve for weight-loss surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged from 18 to 65 years of age, inclusive
* BMI > 40 or BMI > 35 with co-morbidities
* Eligible for weight-loss surgery
* Planned laparoscopic gastric sleeve resections or Roux-en-Y bypass surgery
* Insurance approval status: approved
* Written informed consent

Exclusion Criteria:

* BMI > 55
* Planned two-stage procedures
* Prior bariatric procedures (including gastric banding)
* Serious mental or physical co-morbidities at the discretion of the Investigator
* Insurance approval status: rejected

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as obese and eligible for weight loss surgery (BMI>40; or BMI>35 with co-morbidities) and the following insurance approval status (Kostenubernahmeantrag): approved.
Sampling Method: Non-Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Mann, MD, Principal Investigator — Universitätsklinik Hamburg Eppendorf
Locations (18):
- Germany (18):
  - Krankenhaus Bad Cannstatt, Bad Cannstatt
  - Bundeswehr Krankenhaus Berlin, Berlin
  - Franziskus Hospital Bielefeld, Bielefeld
  - BHV-Reinikenheide, Bremerhaven
  - Amperklinikum Dachau, Dachau
  - Kreiskrankenhaus Emmendingen, Emmendingen
  - Universitätsklinik Hamburg Eppendorf, Hamburg
  - Ev. Krankenhaus Herne, Herne
  - Klinikum Itzehoe, Itzehoe
  - Marienkrankenhaus Kassel, Kassel
  - Krankenhaus Luebbecke, Lübbecke
  - Sana Klinikum Lübeck, Lübeck
  - Diakoniekrankenhaus Mannheim, Mannheim
  - Krankenhaus Hetzelstift Neustadt/Weinstraße, Neustadt
  - Thüringen-Kliniken "Georgius Agricola", Saalfeld
  - Diakonie-Klinikum Schwäbisch Hall, Schwäbisch Hall
  - Schwarzwald Baar Klinikum Villingen, Villingen
  - Krankenhaus Winsen, Winsen

REFERENCES:
- [Derived] Wolter S, Dupree A, ElGammal A, Runkel N, Heimbucher J, Izbicki JR, Mann O, Busch P. Mentorship Programs in Bariatric Surgery Reduce Perioperative Complication Rate at Equal Short-Term Outcome-Results from the OPTIMIZE Trial. Obes Surg. 2019 Jan;29(1):127-136. doi: 10.1007/s11695-018-3495-2. PMID 30187421

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 293 adults were enrolled from 17 Mentor (performed at least 50 procedures) and Mentee (performed less than 50 procedures) bariatric German referral centres. They were stratified for laparoscopic sleeve gastrectomies and Roux en Y gastric bypass (ideally 50:50). First participant enrolled April 2012 Last participant enrolled October 2013.
Pre-assignment Details: Use or preference of surgical procedure was at the discretion of the surgeon. For each patient, the study consisted of three phases: Screening/Baseline; Surgery; Post-operative observation for up to 12 months. Data were gathered per SoC (Standard of Care) at each of the three study phases.
Period: Overall Study
Arm/Group | Procedure Type 1 | Procedure Type 2
Started | 169 | 124
Completed | 117 | 97
Not Completed | 52 | 27
Not completed — Lost to Follow-up | 39 | 14
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Other | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Procedure Type 1 | Procedure Type 2 | Total
Number analyzed (Participants) | 169 | 124 | 293
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 169 | 124 | 293
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 96 | 209
  Male | 56 | 28 | 84
Region of Enrollment [Number; unit: participants]
  Germany | 169 | 124 | 293
Weight (Kgs) [Mean (Standard Deviation); unit: Kgs] | 140.8 (20.6) | 132.3 (20.2) | 137.2 (20.8)
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 47.6 (4.6) | 45.8 (5.0) | 46.8 (4.9)
Type of Insurance (Public/Private) [Number; unit: participants]
  Private Health Insurance | 155 | 119 | 274
  Public Health Insurance | 14 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life (QOL) in First Postoperative Year According to EuroQol-5 Dimensions-5 Levels (EQ-5D-5L)
Description: The EQ-5D-5L (minimum and maximum values are 0 and 1 respectively) consists of two sections,the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).The EQ-5D descriptive system comprises the following five dimensions: mobility,self-care,usual activities (e.g.,work, study..), pain/discomfort and anxiety/depression with five response levels for each dimension:no problems,slight problems, moderate problems,severe problems and extreme problems.The EQ-5D VAS is a 20 cm vertical scale where patients can mark from 0 (worst health imaginable) to 100 (best health imaginable).The global score at each timepoint is calculated as a composite of the five dimention score and of the VAS health score according to a specific algorithm.The Aurea Under the Curve (AUC) of QOL as assessed by EQ-5D-5L is reported to combine repeated measurements at flexible time intervals between 0 and 12 months post-procedure into a single numeric value.The higher the AUC value is,the better the patient is.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: Score*months
Groups:
- Procedure Type I: Gastric Sleeve Resection
- Procedure Type II: Roux-en-Y Gastric Bypass
Arm/Group | Procedure Type I | Procedure Type II
Number analyzed (Participants) | 169 | 124
Score*months | 3 (0.1) | 3 (0.1)

2. Primary Outcome: Quality of Life (QOL) in First Postoperative Year According to Bariatric Analysis and Reporting System (BAROS) With the Moorehead-Ardelt Quality of Life Questionnaire II (M-A QoLQ II)
Description: The BAROS consists of a scoring table that includes three main areas of analysis: weight loss, improvement of medical conditions and M-A QoLQ II. Points are added or subtracted according to changes in these domains. A maximum of three points is given to each domain to evaluate changes after medical or surgical intervention. Points are deducted for complications or reoperations. The M-A QoLQ II assesses six important QoL items (self-esteem, physical activity, social life, work conditions, sexual activity and eating behaviour) on a scale ranging from -0.50 to 0.50 with 0.10 increments to assess each item. The total number of points (range -7 to 9) defines five outcome groups from failure to excellent. The Aurea Under the Curve (AUC) of QOL as assessed by BAROS with M-A QoLQ II is reported to combine repeated measurements at flexible time intervals from 0 to 12 months post-procedure into a single numeric value. The higher the AUC value is, the better the patient is.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Score*months
Arm/Group | Procedure Type 1 | Procedure Type 2
Number analyzed (Participants) | 169 | 124
Score*months | 13 (1.2) | 13 (1.0)

3. Primary Outcome: Quality of Life (QOL) in First Postoperative Year According to Impact of Weight on Quality of Life-Lite Questionnaire (IWQOL-Lite)
Description: The IWQoL-Lite consists of five domains: physical function (11 items), self-esteem (7 items), sexual life (4 items), public distress (5 items), and work (4 items). Each item has five response options: never true-1, rarely true-2, sometimes true-3, usually true-4, and always true-5. In computing raw and normalized scores, a pro-rated system is used for handling missing data. Normalized scores are used to obtain scores ranging from 0 (worst QoL) to 100 (best QoL). The Aurea Under the Curve (AUC) of QOL as assessed by IWQOL-Lite questionnaire is reported to combine repeated measurements at flexible time intervals from 0 to 12 months post-procedure into a single numeric value. The higher the AUC value is, the better the patient is.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Score*months
Arm/Group | Procedure Type 1 | Procedure Type 2
Number analyzed (Participants) | 169 | 124
Score*months | 45 (8.2) | 47 (5.8)

4. Secondary Outcome: Excess Weight Loss (EWL)
Description: EWL, calculated as a percentage, was used to compare weight loss between patients or types of bariatric procedures instead of actual weight loss.
  The formula used was: EWL = 100 × actual weight loss (lbs)/(initial weight [lbs] - IBW [lbs]), where Actual weight loss was calculated as the difference between initial/pre-operative weight (lbs) and post-operative weight (lbs) and IBW was based on the 1983 Metropolitan Height (inches) and Weight (lbs). The Aurea Under the Curve (AUC) of EWL is reported to combine repeated measurements at flexible time intervals from 0 to 12 months post-procedure into a single numeric value. The higher the AUC value is, the more the patient lost weight.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: Percentage EWL*month
Arm/Group | Procedure Type 1 | Procedure Type 2
Number analyzed (Participants) | 169 | 124
Percentage EWL*month | 58 (2.3) | 58 (2.0)

5. Secondary Outcome: Health Resource Utilization - Durantion of Sugery
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Procedure Type 1 | Procedure Type 2
Number analyzed (Participants) | 169 | 124
Minutes | 83.2 (33.5) | 135.9 (51.0)

6. Secondary Outcome: Health Resource Utilization - Recovery Time From Surgery
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Procedure Type 1 | Procedure Type 2
Number analyzed (Participants) | 169 | 124
Days | 7.7 (4.4) | 7.6 (4.1)

7. Secondary Outcome: Health Resource Utilization - Amount of Patients Requiring Transfer to ICU or Other Special Unit During Hospitalization
Time Frame: 12 Months
Measure: Number; unit: percentage of patients
Arm/Group | Procedure Type 1 | Procedure Type 2
Number analyzed (Participants) | 169 | 124
percentage of patients | 50.9 | 51.6

8. Secondary Outcome: Surgical Complications
Description: Incidence of procedural and post-procedural complications through 30 days post-op.
Time Frame: 30 Days
Measure: Number; unit: participants
Arm/Group | Procedure Type 1 | Procedure Type 2
Number analyzed (Participants) | 169 | 124
participants
  Wound infection | 7 | 6
  Disorder of emptying stomach/increased, new reflux | 1 | 6
  Secondary haemorrhage, intra-abdominal | 2 | 4
  Anastomotic leak | 5 | 1
  Dumping syndrome | 4 | 2
  Urinary tract infection | 2 | 2
  Intra-abdominal abscess | 3 | 0
  Diarrhoea | 1 | 2
  Anastomotic stenosis | 2 | 0
  Symptomatic cholelithiasis | 2 | 0
  Others | 9 | 11

ADVERSE EVENTS:
Description: OPTIMIZE Study was an outcome study conducted OUS and designed without specifying which products could be used (standard of care, not necessarily using Covidien products). As per CIP, AEs were not collected during the study (and not differentiated Serious vs other AEs). Complications are categorized as type and number in the Outcome Measure section
Arm/Group | Procedure Type I | Procedure Type II
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No